CLINICAL TRIAL: NCT04646967
Title: A Randomized Control Trial Evaluating Pain Outcomes of Ketorolac Administration in Children Undergoing Circumcision
Brief Title: An Evaluation of Pain Outcomes of Ketorolac Administration in Children Undergoing Circumcision
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alberta Children's Hospital (Other)
Responsible Party: Principal Investigator, Bryce Weber, Pediatric Urologist, Alberta Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REB20-1076
Record Dates: First submitted 2020-11-23; First posted 2020-11-30 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Pain, Postoperative; Phimosis; Paraphimosis; Balanitis
Keywords: penis; pain; ketorolac; circumcision
MeSH Terms: conditions — Pain, Postoperative; Phimosis; Paraphimosis; Balanitis; Pain | interventions — Bupivacaine; Sevoflurane; Acetaminophen; Ibuprofen; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- No ketorolac (Active Comparator): 15 mg/kg oral dose of acetaminophen is administered prior to surgery. General anesthesia will be induced with sevoflurane via facemask. After establishing venous access, a laryngeal mask will be inserted, and anesthesia maintained with 1 minimum alveolar anesthetic concentration (MAC) of sevoflurane in oxygen/air 50/50 mixture. The DPNB nerve block is done using a 23 GA needle inserted below the Buck fascia. Once the needle tip is positioned appropriately and after a negative aspiration test, 0.2mL/kg (maximum 10mL) of 0.25% bupivacaine is injected in small aliquots, with intermittent aspiration throughout. In all patients, skin incision is performed at least 5 min after placement of the nerve block. Patients will be advised to take ibuprofen and acetaminophen postoperatively as needed.
  Interventions: Drug: Bupivacain; Drug: Sevoflurane; Drug: Acetaminophen; Drug: Ibuprofen
- Peri-operative ketorolac (Experimental): Exactly same as the no ketorolac group except at the beginning of the circumcision, once the patient is asleep, patients in the perioperative ketorolac group will also receive a 0.5 mg/kg intravenous dose of ketorolac.
  Interventions: Drug: Bupivacain; Drug: Sevoflurane; Drug: Acetaminophen; Drug: Ibuprofen; Drug: Ketorolac

INTERVENTIONS:
Drug: Bupivacain — See active comparator description
  Other Names: Marcaine
Drug: Sevoflurane — See active comparator description
  Other Names: Sevorane; Ultane; Sojourn
Drug: Acetaminophen — See active comparator description
  Other Names: Tylenol
Drug: Ibuprofen — See active comparator description
  Other Names: Advil
Drug: Ketorolac — See experimental arm description
  Other Names: Toradol
  Arms: Peri-operative ketorolac

SUMMARY:
Circumcision is the most common surgical procedure performed by Pediatric Urologists. Ketorolac has been shown to have an efficacy similar to morphine in multi-modal analgesic regimens without the commonly associated adverse effects. This study aims to see if giving ketorolac during the operation will result in better pain control. We hypothesize that ketorolac will result in pain control similar to morphine with a lower incidence of side effects such as nausea and vomiting.

DETAILED DESCRIPTION:
We performed a pilot study in 2017 evaluating the perioperative use of ketorolac in circumcision. Overall, there were no adverse reactions and ketorolac patients did not experience significantly less pain that the control group patients. However, parental perception of pain was lower in the ketorolac group when compared to the control and this required more investigation. Based on our findings of the pilot study, we determined that we needed at least 36 patients in each study group to come to a statistical conclusion. With a larger study group perhaps a statistical difference in pain as measured with a FLACC score may become apparent.

Prospective, randomized, single-blinded study will be conducted from January 2021 - January 2022. A total of two groups will present with 50 children in each group.

A computer-generated randomized block design program will be used to allocate patients to either the treatment (ketorolac) or control (no ketorolac) group. All children will receive a 15 mg/kg oral dose of acetaminophen prior to surgery unless contraindicated. General anesthesia will be induced with sevoflurane via facemask. After establishing venous access, a laryngeal mask will be inserted, and anesthesia maintained with 1 minimum alveolar anesthetic concentration (MAC) of sevoflurane in oxygen/air 50/50 mixture. The DPNB nerve block will be performed by a pediatric urologist using a 23 GA needle inserted below the Buck fascia. Once the needle tip is positioned appropriately, and after a negative aspiration test, 0.2mL/kg (maximum 10mL) of 0.25% bupivacaine is injected in small aliquots, with intermittent aspiration throughout. In all patients, skin incision is performed at least 5 min after placement of the nerve block. At the beginning of the circumcision procedure once the patient is asleep, patients in the treatment group will receive a 0.5 mg/kg intravenous dose of ketorolac. Patients will be advised to take ibuprofen and acetaminophen post-operatively as needed, but not ibuprofen within 6 hours of the procedure. A 6-hour window between ibuprofen and ketorolac is in line with our standard of practice at the Alberta Children's Hospital when using additional NSAIDs after ketorolac.

Patients' demographic information, time needed to perform the block, time of block onset and duration of surgery will be recorded. The mean arterial pressure, heart rate and oxygen saturation, expired sevoflurane end tidal concentration and MAC will be systematically collected pre-operatively, intra-operatively and post-operatively in the recovery room. The primary outcome of post-operative pain will be evaluated through the use of the Face, Legs, Activity, Cry, Consolability (FLACC) pain score or Numerical Rating Scale (NRS) pain score ascertained by a nurse or research assistant blinded to the anesthetic technique. The usage of these two scales will be performed as deemed appropriate by the research assistant. The FLACC scale will be used in children who have difficulty verbalizing pain and in sleeping children (regardless of age) while the NRS pain score will be used in patients capable of self-assessment (> 7 years of age). The FLACC score is a well-established postoperative pain measure using 5 items scored between 0-2, which has been validated in patients from 6 months up to 7 years of age. These faces are rated on a scale of 10. A FLACC or NRS pain score will be recorded every 15 minutes for the first hour and every 30 minutes for up to 2 hours following discharge from the PACU into the day stay surgical unit. If the score is found to be >3 (moderate pain 4-6, severe pain 7-10), the patient will receive an intravenous morphine dose of 0.05mg/kg. An additional dose may be given 15 minutes following the initial dose of morphine if analgesia is inadequate (score >4). Postoperatively, the child will be monitored every 15 minutes during the first hour and every 30 minutes for the next 2 hours until discharge home. Discharge will be based on normal institutional criteria including level of awareness, hemodynamic stability and absence of pain, bleeding, nausea and vomiting. Prior to discharge, parents will be provided with any additional analgesics required at home and will be contacted 24 hours following their surgery to complete the parents' postoperative pain measure (PPPM). The PPPM is a well-established post-operative pain assessment tool with high inter-rater reliability and construct validity, which has been designed specifically for use by parents in the post-operative care of their children. The measure includes 15 items scored between 0 and 1. The questionnaire will be completed over the telephone at a time corresponding to 24 hours post-surgical closure. Amount of pain and analgesia consumption data will then be collected by contacting the parents 24 hours post procedure.

ELIGIBILITY:
Inclusion Criteria:

* All children admitted for circumcision at the Alberta Children's Hospital

Exclusion Criteria:

* History of allergic reactions to local anesthetics or ketorolac

  * Bleeding diatheses
  * Coagulopathy
  * Infection at the injection site.

Max Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Post-operative pain | Immediately following the procedure
  Evaluated through the use of the Face, Legs, Activity, Cry, Consolability (FLACC) pain score or Numerical Rating Scale (NRS) pain score ascertained by a nurse or research assistant blinded to the anesthetic technique. The FLACC scale will be used in children who have difficulty verbalizing pain and in sleeping children (regardless of age) while the NRS pain score will be used in patients capable of self-assessment.
Post-operative pain | 15 minutes post-operatively
  Evaluated through the use of the Face, Legs, Activity, Cry, Consolability (FLACC) pain score or Numerical Rating Scale (NRS) pain score ascertained by a nurse or research assistant blinded to the anesthetic technique. The FLACC scale will be used in children who have difficulty verbalizing pain and in sleeping children (regardless of age) while the Wong-Baker FACES scale will be used in patients capable of self-assessment. Both scores are out of 10 and can be averaged together to quantify post-operative pain
Post-operative pain | 30 minutes post-operatively
  Evaluated through the use of the Face, Legs, Activity, Cry, Consolability (FLACC) pain score or Numerical Rating Scale (NRS) pain score ascertained by a nurse or research assistant blinded to the anesthetic technique. The FLACC scale will be used in children who have difficulty verbalizing pain and in sleeping children (regardless of age) while the NRS pain score will be used in patients capable of self-assessment.
Post-operative pain | 45 minutes post-operatively
  Evaluated through the use of the Face, Legs, Activity, Cry, Consolability (FLACC) pain score or Numerical Rating Scale (NRS) pain score ascertained by a nurse or research assistant blinded to the anesthetic technique. The FLACC scale will be used in children who have difficulty verbalizing pain and in sleeping children (regardless of age) while the NRS pain score will be used in patients capable of self-assessment.
Post-operative pain | 60 minutes post-operatively
  Evaluated through the use of the Face, Legs, Activity, Cry, Consolability (FLACC) pain score or Numerical Rating Scale (NRS) pain score ascertained by a nurse or research assistant blinded to the anesthetic technique. The FLACC scale will be used in children who have difficulty verbalizing pain and in sleeping children (regardless of age) while the NRS pain score will be used in patients capable of self-assessment.
Post-operative pain | 90 minutes post-operatively
  Evaluated through the use of the Face, Legs, Activity, Cry, Consolability (FLACC) pain score or Numerical Rating Scale (NRS) pain score ascertained by a nurse or research assistant blinded to the anesthetic technique. The FLACC scale will be used in children who have difficulty verbalizing pain and in sleeping children (regardless of age) while the NRS pain score will be used in patients capable of self-assessment.
Post-operative pain | 120 minutes post-operatively
  Evaluated through the use of the Face, Legs, Activity, Cry, Consolability (FLACC) pain score or Numerical Rating Scale (NRS) pain score ascertained by a nurse or research assistant blinded to the anesthetic technique. The FLACC scale will be used in children who have difficulty verbalizing pain and in sleeping children (regardless of age) while the NRS pain score will be used in patients capable of self-assessment.
Post-operative pain | 150 minutes post-operatively
  Evaluated through the use of the Face, Legs, Activity, Cry, Consolability (FLACC) pain score or Numerical Rating Scale (NRS) pain score ascertained by a nurse or research assistant blinded to the anesthetic technique. The FLACC scale will be used in children who have difficulty verbalizing pain and in sleeping children (regardless of age) while the NRS pain score will be used in patients capable of self-assessment.
Post-operative pain | 180 minutes post-operatively
  Evaluated through the use of the Face, Legs, Activity, Cry, Consolability (FLACC) pain score or Numerical Rating Scale (NRS) pain score ascertained by a nurse or research assistant blinded to the anesthetic technique. The FLACC scale will be used in children who have difficulty verbalizing pain and in sleeping children (regardless of age) while the NRS pain score will be used in patients capable of self-assessment.
Post-operative pain | 24 hours post-operatively
  Evaluated through use of Parents' Post-operative Pain Measure (PPPM) completed via telephone follow-up with parent/guardian 24-hours post-operative.

SECONDARY OUTCOMES:
Total ibuprofen consumption | 24 hours post-operatively
  Evaluated and compiled through anesthesia notes, post-operative nursing care notes and parental telephone follow-up
Total acetaminophen consumption | 24 hours post-operatively
  Evaluated and compiled through anesthesia notes, post-operative nursing care notes and parental telephone follow-up
Incidence of bleeding requiring medical attention | Up to 2 weeks
  Bleeding events will be compiled through post-anesthetic care unit, surgical short stay unit, clinic and emergency department notes

CONTACTS AND LOCATIONS:
Overall Officials: Bryce Weber, MD FRCSC, Principal Investigator — Alberta Children's Hospital
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Allan CY, Jacqueline PA, Shubhda JH. Caudal epidural block versus other methods of postoperative pain relief for circumcision in boys. Cochrane Database Syst Rev. 2003;(2):CD003005. doi: 10.1002/14651858.CD003005. PMID 12804449
- [Background] Brady-Fryer B, Wiebe N, Lander JA. Pain relief for neonatal circumcision. Cochrane Database Syst Rev. 2004 Oct 18;2004(4):CD004217. doi: 10.1002/14651858.CD004217.pub2. PMID 15495086
- [Background] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Background] Adler R, Ottaway MS, Gould S. Circumcision: we have heard from the experts; now let's hear from the parents. Pediatrics. 2001 Feb;107(2):E20. doi: 10.1542/peds.107.2.e20. PMID 11158494
- [Background] Sutters KA, Levine JD, Dibble S, Savedra M, Miaskowski C. Analgesic efficacy and safety of single-dose intramuscular ketorolac for postoperative pain management in children following tonsillectomy. Pain. 1995 Apr;61(1):145-153. doi: 10.1016/0304-3959(94)00166-C. PMID 7644238
- [Background] Gunter JB, Varughese AM, Harrington JF, Wittkugel EP, Patankar SS, Matar MM, Lowe EE, Myer CM 3rd, Willging JP. Recovery and complications after tonsillectomy in children: a comparison of ketorolac and morphine. Anesth Analg. 1995 Dec;81(6):1136-41. doi: 10.1097/00000539-199512000-00004. PMID 7486094
- [Background] De Oliveira GS Jr, Agarwal D, Benzon HT. Perioperative single dose ketorolac to prevent postoperative pain: a meta-analysis of randomized trials. Anesth Analg. 2012 Feb;114(2):424-33. doi: 10.1213/ANE.0b013e3182334d68. Epub 2011 Sep 29. PMID 21965355
- [Background] von Baeyer CL, Spagrud LJ. Systematic review of observational (behavioral) measures of pain for children and adolescents aged 3 to 18 years. Pain. 2007 Jan;127(1-2):140-50. doi: 10.1016/j.pain.2006.08.014. Epub 2006 Sep 25. PMID 16996689
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Chambers CT, Hardial J, Craig KD, Court C, Montgomery C. Faces scales for the measurement of postoperative pain intensity in children following minor surgery. Clin J Pain. 2005 May-Jun;21(3):277-85. doi: 10.1097/00002508-200505000-00011. PMID 15818080
- [Background] Chambers CT, Finley AG, McGrath PJ, Walsh TM. The parents' postoperative pain measure: replication and extension to 2-6-year-old children. Pain. 2003 Oct;105(3):437-443. doi: 10.1016/S0304-3959(03)00256-2. PMID 14527704
- [Background] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics 4.4: 287-291, 2005
- See also: Ketorolac compound summary. Pubchem Substance Website. National Center for Biotechnology, US National Library of Medicine — http://pubchem.ncbi.nlm.nih.gov/compound/3826